CLINICAL TRIAL: NCT04687982
Title: Feasibility and Efficacy of Modified Donor Lymphocytes Infusion (CD45RA Negative Selected) After Haploidentical Transplantation With Post-transplantation Cyclophosphamide in Patients With Hematological Malignancies (ONC-2016-002).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONC-2016-002
Record Dates: First submitted 2020-12-10; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Bone Marrow Transplant Infection; Bone Marrow Transplant Complications; Graft Vs Host Disease; Infection; Hematological Malignancy
Keywords: DLI; CD45+; donor lymphocytes infusion; mDLI; haploidentical transplantation; hematological malignancies
MeSH Terms: conditions — Graft vs Host Disease; Infections; Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mDLI infusion (Experimental): The planned number of mDLI is 3.
  1. Day +50 (+/- 7 days) from allogenic transplant, 1st mDLI 5x105CD3+/kg of recipient.
  2. 4-6 weeks after 1st DLI, 2nd mDLI 1x106CD3+/kg of recipient.
  3. 4-6 weeks after 2nd DLI, 3rd mDLI 5x106CD3+/kg of recipient.
  Interventions: Biological: modified donor lymphocytes infusion (mDLI)

INTERVENTIONS:
Biological: modified donor lymphocytes infusion (mDLI) — The planned number of mDLI is 3.
  1. Day +50 (+/- 7 days) from allogenic transplant, 1st mDLI 5x105CD3+/kg of recipient.
  2. 4-6 weeks after 1st DLI, 2nd mDLI 1x106CD3+/kg of recipient.
  3. 4-6 weeks after 2nd DLI, 3rd mDLI 5x106CD3+/kg of recipient.

SUMMARY:
Interventional non-randomized trial. The duration of study will be 47 months.

After haploidentical transplantation, patients without complications, mainly a GVHD ≥ grade 2, will receive mDLI. mDLI consists of donor lymphocytes infusion, harvested by apheresis the day before the day planned for infusion (or up to -7 days) as outpatient basis in the Day Hospital using a cell separator.

The mDLIs preparation will be performed using a CliniMACS® (Miltenyi). A CD45RA-depletion Product LineTM from Miltenyi, including disposable reagents and devices, will be used.

The planned number of mDLI is 3.

1. Day +50 (+/- 7 days) from allogenic transplant, 1st mDLI 5x105CD3+/kg of recipient.
2. 4-6 weeks after 1st DLI, 2nd mDLI 1x106CD3+/kg of recipient.
3. 4-6 weeks after 2nd DLI, 3rd mDLI 5x106CD3+/kg of recipient. Day +50 was chosen as the starting time-point because at that time over two thirds of all acute GvHD episodes have already occurred in the absence of DLI (internal data, median +49 after bone marrow, +27 after peripheral stem cells); acute GvHD will thus be less likely a confounding factor. The choice of a maximum number of 3 mDLIs is based on the relatively narrow time interval where outcome improvement is expected, that is mainly in the first 6 months after haplo-HSCT. The planned doses are those mainly used in conventional DLIs during haplo-HSCT setting.

Stopping infusion rules:

If GvHD ≥ Grade 2 or relapse occurs, mDLIs will not be administered at any time and patient will be permanently discontinued from treatment.

If any severe adverse event (SAE) occurs after the first mDLI, the administration of mDLI will be interrupted for a maximum of 6 weeks until event resolution. If the SAE does not resolve after 6 weeks from last mDLI infusion, patient will be permanently discontinued. At any time, the experimental treatment may be stopped according to clinical judgement or patient's willing.

ELIGIBILITY:
Inclusion Criteria:

1. Written, signed informed consent;
2. Adult patients aged ≥18 years;
3. Patients who underwent haploidentical transplantation with PT-Cy for haematological diseases since no more than 56 days;
4. Patient who received myeloablative conditioning regimen, reduced intensity conditioning regimens, or non-myeloablative conditioning regimens;
5. Availability of haploidentical donor (defined as those with ≥ 2 differences within one HLA haplotype) who agree to donate peripheral blood cells by leukapheresis and able to donate the day before the day planned for infusion (or up to - 7 days);
6. GVHD/HVG prophylaxis consists in Cyclophosphamide: 50 mg/kg/day, day +3 and +4, Cyclosporine A: 3 mg/kg/day from day +5 to day +100, with tapering in 2 months Mycophenolate mofetil: 45 mg/kg/day, from day +5 to day +35.

Exclusion Criteria:

1. Presence of grade 2-4 acute GVHD;
2. Uncontrolled bacterial, viral or fungal infection;
3. Aplasia defined as ANC less than 500/L;
4. Evidence of disease progression after transplantation;
5. Current participation in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
to evaluate the efficacy of CD45RA-depleted haplo-DLIs (mDLIs) in the setting of patients receiving haplo-HSCT and PT-Cy, in terms of incidence of viral infections in the post-transplant period | 100 days
  The primary endpoint is the rate of viral infections at day +100 after haplo-BMT.
to evaluate the impact of the modified DLIs on the occurrence of GvHD | 1 year
  acute and chronic GvHD incidence
to evaluate the impact of the modified DLIs on relapse (graft-versus-tumor effect) | 1 year
  relapse rate
to evaluate the impact of the modified DLIs on other types of infections; | 100 days
  100-day cumulative incidence of other type of infections

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Beek JJP, Puccio S, Di Vito C, De Paoli F, Zaghi E, Calvi M, Scarpa A, Peano C, Basso G, Cibella J, De Philippis C, Sarina B, Timofeeva I, Capizzuto R, Mannina D, Mineri R, Mariotti J, Crocchiolo R, Santoro A, Castagna L, Bramanti S, Mavilio D, Lugli E. Selected memory T cells infused post-haploidentical hematopoietic stem cell transplantation persist and hyperexpand. Blood Adv. 2023 Jul 25;7(14):3458-3468. doi: 10.1182/bloodadvances.2022007735. PMID 36469095